CLINICAL TRIAL: NCT06381063
Title: Effect of Non-steroidal Anti-inflammatory Drugs in Pain Management After Cardiac Surgery
Brief Title: Non-steroidal Anti-inflammatory in Cardiac Surgery
Acronym: KETOPAIN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: University Hospital, Rouen (Other); University Hospital, Lille (Other); University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI2023_843_0152
Record Dates: First submitted 2024-04-05; First posted 2024-04-24 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Acute Postoperative Pain; Non-steroidal Anti-inflammatory Drugs; Cardiac Surgery; Pain Intensity; Multimodal Pain Management
Keywords: Acute Postoperative Pain; non-steroidal anti-inflammatory drugs; cardiac surgery; pain intensity; multimodal pain management
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Pain Management; Ketoprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketoprofen (Experimental): Ketoprofen 100 mg twice a day, during 48 after surgery, intravenous administration
  Interventions: Drug: pain management; Drug: ketoprofen
- Placebo (Placebo Comparator): Placebo twice a day, during 48 h after surgery, intravenous administration
  Interventions: Drug: pain management; Drug: PLacebo

INTERVENTIONS:
Drug: pain management — o Pain management in both arms Intraoperative time: intravenous ketamine 0.5 mg kg-1, intravenous dexamethasone 8 mg Postoperative time: paracetamol 1 g every 6 hours a day, nefopam 20 every 8 hours a day, patient control analgesia with morphine or oxycontin
Drug: ketoprofen — Ketoprofen 100 mg twice a day, during 48 after surgery, intravenous administration
  Arms: Ketoprofen
Drug: PLacebo — Placebo twice a day, during 48 h after surgery, intravenous administration
  Arms: Placebo

SUMMARY:
Non-steroidal anti-inflammatory drugs (NSAID) are part the multimodal strategy in pain management after surgery. However, major concerns are raised in cardiac surgery given the potential side effects of NSAID with more bleeding and acute kidney injury. The investigators hypothesized that NSAID are safe in the early postoperative course after cardiac surgery with respect to contraindication.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for cardiac surgery (aortic valve replacement, coronary artery bypass graft, mitral valve repair or replacement, intracardiac tumor, aortic root repair)
* under cardiopulmonary bypass
* Affiliation to the French national healthcare system
* Written consent obtained

Exclusion Criteria:

* age<18
* weight<50 kg
* chronic use of NSAID
* mini-invasive surgery
* NSAID contraindication
* NSAID allergy
* Nefopam contraindication
* Paracetamol contraindication
* Tramadol contraindication
* Urgent surgery
* Endocarditis
* Immunosuppressive drug
* HIV infection with CD4<200 mm3
* Organ transplantation
* Stage 4 or 5 chronic kidney disease
* Gastro duodenal ulcer
* Pregnancy
* Depression
* Auto immune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
reduction in pain intensity during chest physiotherapy at 24 hours from the end of surgery | at 24 hours
  Pain intensity will be assessed using the NRS at 24 hours from the end of surgery during chest physiotherapy
NSAIDs reduce postoperative at rest at 24 hours from the end of surgery | at 24 hours
  Pain intensity will be assessed at rest at 24 hours from the end surgery using the numerous rating scale (NRS) graded from 1 (no pain) to 10 (high pain intensity)

SECONDARY OUTCOMES:
Change in pain trajectory during the first 7 days after cardiac surgery | 7 days
  Pain trajectory will be assessed every day using NRS and trajectory will be defined as following
Change in cumulative opioid within 48 hours after surgery | 48 hours
  Total dose of oxynorm or morphine will be recorded from the end of surgery to 48 h after and expressed in milligram
Change in pulmonary postoperative complications within 7 days after surgery | 7 days
  Postoperative pulmonary complications will be defined by the occurrence of at least one item among following: atelectasis, pneumonia, acute respiratory distress syndrome, acute respiratory failure, bronchospasm

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huette P, Moussa M, Diouf M, Lefebvre T, Bayart G, Guilbart M, Viart C, Haye G, Bar S, Caus T, Soriot-Thomas S, Boddaert S, Alshatri HY, Tarpin P, Fumery O, Beyls C, Dupont H, Mahjoub Y, Besnier E, Abou-Arab O. Effect of non-steroidal anti-inflammatory drugs on the management of postoperative pain after cardiac surgery: a multicenter, randomized, controlled, double-blind trial (KETOPAIN Study). Trials. 2024 Sep 16;25(1):613. doi: 10.1186/s13063-024-08326-z. PMID 39285437